CLINICAL TRIAL: NCT02601274
Title: Open-label, Dose Escalation Phase I Study of Theliatinib (HMPL-309,Xiliertinib) in Patients With Advanced Solid Tumors
Brief Title: Study of Theliatinib (HMPL-309) in Patients With Advanced Solid Tumor
Acronym: HMPL-309
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: the change of clinical development plan
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-309-00CH1
Record Dates: First submitted 2015-10-20; First posted 2015-11-10 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group Assignment (Experimental): Theliatinib investigational product once a day (QD) will be orally administrated on a 28-day cycle There are 7 dose cohorts,including120mg/160mg/200mg/220mg/300mg/400mg/500mg, QD in the dose escalation stage .
  Interventions: Drug: Theliatinib

INTERVENTIONS:
Drug: Theliatinib — Theliatinib is a tablet in the form of 25 mg ,10mg and 100 mg,oral,once daily
  Other Names: HMPL-309,xiliertinib

SUMMARY:
A Phase I, open-label, multicenter dose-escalation study to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of hmpl-309 in patients with advanced solid tumors

DETAILED DESCRIPTION:
There are two stages to this study: a dose-escalation stage and a dose-expansion stage.

Dose-escalation stage: hmpl-309 administered orally once every day(QD) to patients with locally advanced or metastatic solid tumors for whom standard therapy either does not exist or has proven to be ineffective or intolerable. Dose-expansion stage: hmpl-309 administered orally 300mg once every day(QD) to patients which is only for patients with EGFR positive oesophageal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology confirmed solid tumors
* Failed to standard treatment or no standard treatments for uncontrolled, recurrent and/or metastatic advance tumor (whatever previous surgery conditions)

Dose-escalation stage:

<300mg/day cohort no requiremnet for pathological pattern >300mg/day cohort required NCSLC, head and net squamous carcinoma, or oesophageal carcinoma Dose-expansion stage required oesophageal carcinoma

* Age 18-75
* performance status of 0, or 1, and no worse within 7days
* Life expected >3 months
* written informed consent form voluntarily

Exclusion Criteria:

* Lab testing within 1 week before enrolled, hemoglobin <9 g/dL or , platelet count < 750,000/mm3 and<150000/mm3,
* Total bilirubin≥1.5× the upper limit of normal,
* Serum creatinine higher than normal range
* Diastolic pressure≥150mmHg or systolic pressure≥100mmHg whatever anti-hypertension drug used,
* Serum potassium (whenever potassium implemented) , serum calcium(ionic or albumin-type calcium) or serum magnesium outside normal ranges(whenever implemented)
* Within previous 4 weeks treated by systemic anti-tumor therapy, or radiotherapy, immune therapy, biological or hormonal therapy, and clinical trials. But exclude the below therapy, Prostate cancer treated by hormonal therapy such as GnRH(gonadotropin-releasing hormone) analogue or antagonist Hormone replacement therapy or oral contraceptive Palliative radiotherapy for bone metastasis within 2 weeks
* Prior documental evidence of resistance to EGFR-TKI (epidermal growth factor receptor-tyrosine kinase inhibitors)
* Unrecovered from any previous therapy related toxicity to≤ CTCAE(Common Toxicity Criteria for Adverse Effects) 0 or 1or unrecovered from any previous surgery
* Any CNS(central nervous system) metastasis with uncontrolled symptoms
* Known dysphagia or drug malabsorption
* Active infections such as acute pneumonia, hepatitis B active period
* APTT (activated partial thromboplastin time) and/or INR(international normalized ratio), PT≥2 the upper limit of normal(not including patients treated by anticoagulation treatment)
* ocular surface diseases or dry eye syndrome
* skin disease with obvious symptoms and signs
* significant cardiovascular disease, including II-IV atrioventricular block, acute myocardial infarction within 6 months, significant angina or Coronary artery bypass graft
* Known existing interstitial lung disease
* Female patients who are pregnant or feeding, or childbearing potential patient with pregnant testing positive
* Any abnormal of clinical and laboratory so that patients unsuitable to attend the trial sine in the opinion of the investigator
* Patients unable to comply with the protocol since significant psychological or psychogenic abnormal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
incidence of all types/grades of adverse events | from first patient in till 30 days after the last patient last visit
  for each patient, adverse events are collected from the date of consent until 30 days after trial discontinuation

OTHER OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Day 1-3 Single Dose and Day 1-28 Steady State
  Based on single-dose PK result, multi-dose stage subjects take HMPL-309 once a day or twice a day, PK samples are collected of a single oral dose of HMPL-309 on Day 1 to Day 3. At multiple-dose, Pharmacokinetics(PK) sampling will include a pre-dose and at the 0.5,2,4,6,8 hour time points on days 1,15,21of dosing in the first 21-Day cycle of therapy, and pre-dose on days 2,8,16,and 22 of the first 21-Day cycle of therapy
Peak Plasma Concentration (Cmax) | Day 1-3 Single Dose and Day 1-28 Steady State
  Based on single-dose PK result, multi-dose stage subjects take HMPL-309 once a day or twice a day, PK samples are collected of a single oral dose of HMPL-309 on Day 1 to Day 3. At multiple-dose, Pharmacokinetics(PK) sampling will include a pre-dose and at the 0.5,2,4,6,8 hour time points on days 1,15,21of dosing in the first 21-Day cycle of therapy, and pre-dose on days 2,8,16,and 22 of the first 21-Day cycle of therapy

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun-Yat-sen univercity cancer centre, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No